CLINICAL TRIAL: NCT01520714
Title: Effect of Posture on LV Transvenous Lead Capture Thresholds (EXPECT)
Brief Title: Effect of Posture on Left Ventricular (LV) Transvenous Lead Capture Thresholds (EXPECT)
Acronym: EXPECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower enrollment rate than expected
Sponsor: Baylor Research Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 009-067
Record Dates: First submitted 2010-02-22; First posted 2012-01-30 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure (CHF); Cardiac Resynchronization Therapy (CRT); BiVentricular Implantable Cardioverter Defibrillator (BiVICD); Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medtronic passive fixation LV lead (Experimental): Medtronic 4195 Active Fixation LV lead and Medtronic passive fixation LV lead arms will both have same follow-up testing and schedule
  Interventions: Device: Medtronic 4195 active fixation LV lead and Medtronic passive fixation LV lead
- Medtronic 4195 Active Fixation LV Lead (Experimental): Medtronic 4195 Active Fixation LV lead and Medtronic passive fixation LV lead arms will both have same follow-up testing and schedule
  Interventions: Device: Medtronic 4195 active fixation LV lead and Medtronic passive fixation LV lead

INTERVENTIONS:
Device: Medtronic 4195 active fixation LV lead and Medtronic passive fixation LV lead — 1:1 randomization between Medtronic active fixation 4195 LV lead and another FDA approved passive fixation Medtronic LV lead. Fluoroscopic images will be taken at implant in a supine position and again at 3 month follow-up in different postural positions with capture thresholds of the LV lead taken at each postural position.

SUMMARY:
The purpose of this study is to determine whether changes in a patient's position affect LV capture thresholds in a clinically significant way.

DETAILED DESCRIPTION:
Traditionally clinicians program the safety margins for the right atrial, right ventricular, and left ventricular leads two-times the capture thresholds. This safety margin is necessary for the right atrial and right ventricular outputs to prevent asystole during fluctuation of capture thresholds. This two-times safety margin may not be necessary for the left ventricular lead output and may be causing shorter device battery longevity. Newly implemented LV capture threshold management algorithms may help maintain a proper balance of safety margin and battery longevity. However, recent research conducted on automatic left ventricular capture measurement (LVCM) shows as much as 3.5 V daily variability in capture thresholds. In this same study, 18% of patients had >1.5 V LV threshold variability. A possible explanation for the variability of LV thresholds is lead stability. Small movements of the lead electrodes associated with movement of patient posture may account for daily fluctuation of capture thresholds. As heart failure patient care and therapies improve, CRT patients may survive longer than the projected longevities of their device. In order to minimize patient risks associated with device change-outs, care must be taken to maximize battery longevity while maintaining CRT pacing. Examining patient posture changes as a possible cause of threshold variability may guide clinicians to program more appropriate LV outputs with patient safety and device longevity in mind.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age and able to provide informed consent
* Planned placement of a Medtronic LV pacing lead and a Medtronic ICD generator with LVCM technology
* Geographically stable and able to follow-up for a period of at least six months post-procedure at The Heart Hospital Baylor Plano
* Willingness to comply with the requirements of the protocol

Exclusion Criteria:

* Life expectancy of less than six months
* Plans for or significant possibility of pregnancy during the required follow-up window
* Significant cardiovascular surgery planned within six months following ICD implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B DeVille, M.D., Principal Investigator — Baylor Research Institute - The Heart Hospital Baylor Plano
Locations (1):
- The Heart Hospital in Plano, Plano, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients required at physician office. Recruiting will be active until 40 patients are randomized.
Groups:
- Medtronic Passive Fixation LV Lead; Medtronic 4195 Active Fixation LV Lead: Medtronic 4195 Active Fixation LV lead and Medtronic passive fixation LV lead arms will both have same follow-up testing and schedule
  Medtronic 4195 active fixation LV lead and Medtronic passive fixation LV lead : 1:1 randomization between Medtronic active fixation 4195 LV lead and another FDA approved passive fixation Medtronic LV lead. Fluoroscopic images will be taken at implant in a supine position and again at 3 month follow-up in different postural positions with capture thresholds of the LV lead taken at each postural position.
Period: Overall Study
Arm/Group | Medtronic Passive Fixation LV Lead | Medtronic 4195 Active Fixation LV Lead
Started | 0 | 11
Completed | 0 | 5
Not Completed | 0 | 6
Not completed — Protocol Violation | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medtronic Passive Fixation LV Lead | Medtronic 4195 Active Fixation LV Lead | Total
Number analyzed (Participants) | 0 | 11 | 11
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 7 | 7
  >=65 years |  | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 65 (11) | 65 (11)
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 10 | 10
Region of Enrollment [Number; unit: participants]
  United States |  | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Change in Threshold of >1 Volt With Posture Changes
Time Frame: 6 months
Population: Early termination leading to small numbers of subjects; Non-efficacy of treatment leading to no data summary and analysis.
Groups:
- Medtronic Passive Fixation LV Lead; Medtronic 4195 Active Fixation LV Lead: Medtronic 4195 Active Fixation LV lead and Medtronic passive fixation LV lead arms both had same follow-up testing and schedule.
  Medtronic 4195 active fixation LV lead and Medtronic passive fixation LV lead: 1:1 randomization between Medtronic active fixation 4195 LV lead and another FDA approved passive fixation Medtronic LV lead. Fluoroscopic images were taken at implant in a supine position and again at 3 month follow-up in different postural positions with capture thresholds of the LV lead taken at each postural position.
Arm/Group | Medtronic Passive Fixation LV Lead | Medtronic 4195 Active Fixation LV Lead
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medtronic 4195 Active Fixation LV Lead | Medtronic Passive Fixation LV Lead
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic 4195 Active Fixation LV Lead (N=11) | Medtronic Passive Fixation LV Lead (N=0)
Pre-existing AF-AVNode ABL (Cardiac disorders) | 1 (1) | 0 (0)
Enteroccoccal Septicemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LV lead dislodgement (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects; Non-efficacy of treatment leading to no data summary and analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No